CLINICAL TRIAL: NCT06538285
Title: Pilot Clinical Trial of Ketamine-assisted Psychotherapy for Methamphetamine Use Disorder and HIV Risk Reduction
Brief Title: Ketamine-Assisted Recovery for Methamphetamine Use Disorder & HIV
Acronym: KARE
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Nicky Mehtani, MD, MPH (Other)
Collaborators: San Francisco Department of Public Health (Other Government); California HIV/AIDS Research Program (Other); National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Sponsor-Investigator, Nicky Mehtani, MD, MPH, Assistant Professor, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H24SB7788; 2KL2TR001870 (NIH)
Record Dates: First submitted 2024-07-31; First posted 2024-08-05 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-02

CONDITIONS: Methamphetamine Use Disorder
Keywords: HIV; Methamphetamine withdrawal; Ketamine-assisted therapy; Psychedelic; Sexual Behavior; Methamphetamine; Ketamine-assisted psychotherapy; Chemsex
MeSH Terms: conditions — Sexual Behavior; Chemsex | interventions — Ketamine; Psychotherapy; Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Ketamine-Assisted Psychotherapy (Experimental): Participants will receive 3 administrations of intramuscular (IM) ketamine, dosed approximately once weekly, in combination with 7 psychotherapy visits over a 5-week treatment period. All ketamine dosing and psychotherapy visits will be conducted in-person in a designated therapy room.
  Interventions: Drug: Ketamine; Behavioral: Psychotherapy

INTERVENTIONS:
Drug: Ketamine — Ketamine 0.50 mg/kg IM will be administered during the first dosing visit, and either 0.50 mg/kg IM or 0.75 mg/kg IM will be administered at the two subsequent dosing visits, depending on the participant's toleration of prior ketamine dose(s). All ketamine dosing visits will be facilitated by a licensed study therapist and clinician (i.e., NP or MD).
  Other Names: Ketalar; Ketamine hydrochloride; Ketamine injection
Behavioral: Psychotherapy — Psychotherapy will consist of three 1-hour preparatory talk therapy sessions over the 14 days preceding the first ketamine dosing visit, a 1-hour integration talk therapy session within 1-3 days following each ketamine dosing visit, and a final 1-hour integration talk therapy session about 1 week following the last ketamine visit. All talk therapy visits will be conducted by a licensed study therapist.
  Other Names: Talk therapy; Therapy

SUMMARY:
The goal of this clinical trial is to learn whether it is possible to use intramuscular (IM) ketamine in combination with psychotherapy to treat moderate-to-severe methamphetamine use disorder (MeUD) in publicly insured patients with or at-risk for HIV disease. The main questions it aims to answer are:

* Do publicly insured patients find ketamine-assisted psychotherapy feasible and acceptable as a potential treatment for MeUD?
* Is IM ketamine safe and tolerable among patients with MeUD?

Participants will:

* Receive 3 monitored doses of IM ketamine
* Have 3 preparation and 4 integration psychotherapy visits
* Report their daily amounts of methamphetamine used prior to, during, and up to 3 months following the intervention

DETAILED DESCRIPTION:
This is a single-arm pilot feasibility trial (N=12) of 3 doses of ketamine hydrochloride (0.50-0.75 mg/kg IM) administered approximately once weekly, in combination with 7 sessions of manualized psychotherapy for publicly insured patients with moderate-to-severe methamphetamine use disorder (MeUD) who have or are at-risk for HIV. Participants will be administered 3 preparatory psychotherapy visits over the 14 days prior to their first ketamine visit, a psychotherapy integration visit within 1-3 days following each ketamine visit, and a final integration visit about 1 week following their last ketamine visit. This 10-visit Ketamine-Assisted Psychotherapy (KAP) treatment intervention will last about 5 weeks in duration, and 2 follow-up assessment visits will be conducted at 4 and 12 weeks following KAP.

Participants will receive ketamine 0.50 mg/kg IM during their initial dosing visit, and either ketamine 0.50 mg/kg IM or 0.75 mg/kg IM at each subsequent dosing visit, depending on their toleration of prior dose(s).

Screening data will be reviewed to determine subject eligibility. Subjects who meet all inclusion criteria and none of the exclusion criteria will be entered into the study.

Evaluations will be taken at baseline and each of the study visits.

The total duration of subject participation will be up to 119 days-including 5 weeks (i.e., 35 days) for the KAP intervention with follow-up assessment visits at 4 weeks (i.e., 28 days) and 12 weeks (i.e., 84 days) post-intervention.

The total duration of the study is expected to be 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-69
* Moderate or severe methamphetamine use disorder
* Interest in reducing or stopping methamphetamine use
* Insured by MediCal, MediCare, or Healthy San Francisco
* Used methamphetamine ≥7 out of the 30 days prior to screening OR enrolled in a residential drug treatment program
* Have a diagnosis of HIV OR taken PrEP over the last 90 days OR engaged in ≥1 risk behavior for HIV acquisition/transmission over the last 90 days (i.e., anal sex under the influence of methamphetamine, condomless sex with a partner of serodiscordant or unknown HIV status, or any shared use of injection drug supplies)
* English speaking
* Permanently housed for ≥30 days OR enrolled in residential drug treatment for ≥5 days
* Have a text-capable cell phone or access to email (if not enrolled in residential treatment)
* Able and willing to provide informed consent and adhere to visit schedule
* If necessary, willing to be contacted on a daily basis by one of the therapists for 7 days after each ketamine session
* Prior to scheduled ketamine sessions, agree: (a) abstain from using methamphetamine and cocaine for ≥48 hours, (b) abstain from using non-prescribed opioids, cannabis products, benzodiazepines, or alcohol for ≥24 hours, (c) consume no more than a modest quantity (e.g., 1 cup) of caffeine (e.g., coffee or tea) in the morning; (d) continue usual regimen of routinely prescribed opioid-based medications throughout trial; and (e) continue any routine behavioral or pharmacologic mental health interventions as usual outside of the trial
* Female-born participants of child-bearing potential with male-born partners and male-born participants with female-born partners of child-bearing potential must agree to use highly effective contraception for at least 1 month prior to and 2 months after ketamine administration

Exclusion Criteria:

* Significant prior use of ketamine for non-anesthetic purposes, as determined by the investigators
* Cognitive impairment sufficient to impede the ability to complete study tasks
* Lifetime history of intracranial hemorrhage
* Has an intracranial mass
* Had a stroke in the past 12 months
* Had a seizure in the past 6 months
* Has current psychosis or any lifetime history of schizophrenia or schizoaffective disorder
* Engaged in a contingency management program during study
* Taking any prohibited medications
* If receiving any medication that may cause blunting of responses or diminished affect, such as antipsychotics, exclusion will be as per the evaluation of the PI and study staff
* Active suicidal ideation with intent
* Baseline hypertension (≥150 SBP or ≥90 DBP) after repeated measurements
* History of aneurysmal vascular disease, dissection or arteriovenous malformation
* Had a cardiac arrest or myocardial infarction in the past 12 months
* QTc >450 msec on 12-lead EKG (Bazett's formula)
* Has a clinically significant arrhythmia
* Meets any of the following laboratory parameters: ALT ≥3x ULN, AST ≥3x ULN, total bilirubin ≥1.5x ULN, eGFR <30mL/min by CKD-EPI or currently on dialysis
* Pregnant, breastfeeding, or unwilling to use birth control during the study
* Pending legal proceedings with a high risk for incarceration during the study
* Taken another investigational drug in the past 30 days
* Has any physical or mental health condition which, per the clinical judgment of the investigators, interferes with safe study participation or adherence to study procedures

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-03-04 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Trial Recruitment | Up to 28 days
  Binary trial feasibility outcome of whether prospective participants undergoing in-person screening (V0) are found to be fully eligible and ultimately enroll in the study (V1).
Trial Completion | Up to 35 days
  Binary trial feasibility outcome of whether enrolled participants complete at least 70% of KAP intervention visits (i.e., Visits #1-10)
Acceptability Questionnaire | Up to 35 days
  At the end of the KAP intervention (i.e., V10), participants will be administered an 8-item, 5-point-scale questionnaire based off of the Sekhon Theoretical Framework of Acceptability to evaluate eight distinct aspects of the acceptability of the intervention. Higher scores indicate greater levels of intervention acceptability.

SECONDARY OUTCOMES:
Adverse Events | Up to 119 days
  Information regarding occurrence of adverse events will be captured throughout the study at every visit (i.e., V1-V12). Duration (start and stop dates), severity/grade, outcome, treatment and relation to study drug will be recorded.
Blood Pressure | Up to 28 days
  During ketamine administration visits (i.e, V4, V6, and V8), blood pressure (in mmHg) will be monitored at serial 15-minute intervals for 60 minutes following ketamine dosing, and subsequently at 30-minute intervals until the session is complete.
Heart Rate | Up to 28 days
  During ketamine administration visits (i.e, V4, V6, and V8), heart rate (in beats per minute) will be monitored at serial 15-minute intervals for 60 minutes following ketamine dosing, and subsequently at 30-minute intervals until the session is complete.
Methamphetamine Use by Timeline Follow Back | Up to 119 days
  The TLFB is a semi-structured interview that provides estimates of the daily quantity, frequency, and pattern of substance use during a specified time period. It uses a calendar prompt and number of other memory aids (e.g., holidays, payday, and other personally relevant dates) to facilitate accurate recall of drug use during the target period. The TLFB has shown adequate to excellent reliability and validity over a wide range of research and clinical contexts. Non-study SUD treatment utilization will also be recorded on the TLFB form.
Methamphetamine Cravings | Up to 119 days
  A Visual Analog Scale (ranging from 0 to 100) will be used to assess participants' overall cravings for methamphetamine at every study visit.
Amphetamine Cessation Symptom Assessment | Up to 119 days
  The ACSA is a 16-item, 5-point scale (0 = "Not at all" to 4 "Extremely") measuring various aspects of anxiety and mood, fatigue, and craving to measure the severity of amphetamine withdrawal symptoms over the past 24 hours. Higher scores reflect more severe withdrawal symptoms. The ACSA will be administered at all non-ketamine dosing visits (i.e., V1-V3, V5, V7, V9-V12).
Methamphetamine Positive Urine Drug Screens | Up to 119 days
  A point-of-care urine drug screen (UDS) will be collected at every study visit (i.e., V1-V12).
Methamphetamine Levels in Hair | Up to 119 days
  At baseline (V1), end-of-treatment (V10) and 4- and 12-weeks follow-up (V11 and V12), a 1-cm hair sample will be collected from the back of the scalp to measure cumulative drug levels of methamphetamine over the preceding one month period. Quantification of methamphetamine levels in hair will each require a sample of 50-100 strands, which is roughly the equivalent to the average amount of natural hair loss that occurs on a daily basis.
Antiretroviral Adherence | Up to 119 days
  If applicable, self-reported days of antiretroviral drug adherence will be measured at baseline (i.e., V1), end-of-treatment (V10), and at 4- and 12-weeks post-KAP (i.e., V11 and V12).
Depression Symptoms | Up to 119 days
  The Patient Health Questionnaire-9 (PHQ-9) is a validated and widely-used 9-item, 4-point scale (0 = "Not at all" to 3 = "Nearly every day") that assesses depression symptom severity with a 2-week recall period. Higher scores indicate worse depression. It will be administered at baseline (V1), mid-KAP (V7), end-of-treatment (V10), and at 4- and 12-weeks post-KAP (i.e., V11 and V12).
Anxiety Symptoms | Up to 119 days
  The (GAD-7) is a validated self-report measure for the severity of generalized anxiety disorder (GAD) symptoms. This 7-item, 4-point scale (0 = "Not at all" to "3 = Nearly every day") scale has 2-week recall period. Item scores are summed to produce a total score that can range 0-21, with higher scores indicating greater severity of symptoms of GAD.
  It will be administered at baseline (V1), mid-KAP (V7), end-of-treatment (V10), and at 4- and 12-weeks post-KAP (i.e., V11 and V12).

OTHER OUTCOMES:
Attachment Insecurity | Up to 119 days
  The Experiences in Close Relationships - Revised Questionnaire (ECR-R) is a 36-item measure of adult attachment style that measures individuals on two 18-item subscales of attachment: Avoidance and Anxiety. Higher scores on each subscale indicate higher levels of avoidance or anxiety in close relationships. Attachment insecurity has been highly correlated with substance use and changes in the severity of attachment insecurity may underly changes in addictive behaviors. The ECR-R will be administered at baseline (V1), following the last ketamine administration (V9), and at 4- and 12-weeks post-KAP (i.e., V11 and V12).

CONTACTS AND LOCATIONS:
Overall Officials: Nicky Mehtani, MD MPH, Principal Investigator — University of California, San Francisco
Locations (1):
- San Francisco Department of Public Health, San Francicso, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mehtani NJ, Anderson BT, Alexander I, Hendricks PS, Mitchell JM, Coffin PO, Johnson MO. Ketamine-Assisted Recovery (KARE): protocol for an open-label pilot trial of ketamine-assisted psychotherapy for publicly insured patients with methamphetamine use disorder and HIV risks. BMJ Open. 2025 Aug 24;15(8):e100775. doi: 10.1136/bmjopen-2025-100775. PMID 40850924